CLINICAL TRIAL: NCT03960138
Title: Examining the Effects of Theta Burst Stimulation on Corticothalamic Mediated Inhibitory Control and Smoking Relapse Vulnerability
Brief Title: Examining the Effects of Neural Stimulation on Inhibitory Control and Cigarette Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Brett Froeliger, Professor Psychiatry, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 00074836
Record Dates: First submitted 2019-05-10; First posted 2019-05-22 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intermittent Theta-burst stimulation (iTBS) (Experimental): Cross-over design - participants will receive both experimental treatments.
  Interventions: Device: Intermittent Theta-burst stimulation (iTBS); Device: Continuous Theta-burst stimulation (cTBS)
- Continuous Theta-burst stimulation (cTBS) (Experimental): Cross-over design - participants will receive both experimental treatments.
  Interventions: Device: Intermittent Theta-burst stimulation (iTBS); Device: Continuous Theta-burst stimulation (cTBS)

INTERVENTIONS:
Device: Intermittent Theta-burst stimulation (iTBS) — Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected.
Device: Continuous Theta-burst stimulation (cTBS) — Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Continuous TBS (cTBS) which is thought to temporarily dampen brain activity in that specific area.

SUMMARY:
The purpose of this research study is to examine the effects of theta-burst Transcranial Magnetic Stimulation on inhibitory control and smoking among adult cigarette smokers.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 18 and 65.
2. Be in stable mental and physical health.
3. Be willing to provide informed consent.
4. Be able to comply with protocol requirements and likely to complete all study procedures.
5. Be a current nicotine dependent cigarette smoker (smoke ≥10 cigs/day) with a minimum smoking history of smoking an average of ≥ 10 cigs/day over the past two years.

Exclusion Criteria:

* 1. Contraindication to MRI (e.g., presence of metal in the skull, orbits or intracranial cavity, claustrophobia).

  2. Contraindication to TMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for > 15 minutes, implanted electronic device, metal in the head, or pregnancy, as indicated by a positive urine pregnancy test at screening).

  3. Any use of substances that lower seizure threshold (such as thyroid medications or cocaine).

  4. History of autoimmune, endocrine, viral, or vascular disorder affecting the brain.

  5. History or MRI evidence of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment.

  6. Unstable cardiac disease, uncontrolled hypertension, severe renal or liver insufficiency, or sleep apnea.

  7. BAC greater than 0.0. 8. Any other condition or concern that in the Investigator's opinion would impact participant safety, compliance with study instructions, or potentially confound the interpretation of the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri - Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Froeliger B, McConnell PA, Bell S, Sweitzer M, Kozink RV, Eichberg C, Hallyburton M, Kaiser N, Gray KM, McClernon FJ. Association Between Baseline Corticothalamic-Mediated Inhibitory Control and Smoking Relapse Vulnerability. JAMA Psychiatry. 2017 Apr 1;74(4):379-386. doi: 10.1001/jamapsychiatry.2017.0017. PMID 28249070
- [Derived] Upton S, Brown AA, Ithman M, Newman-Norlund R, Sahlem G, Prisciandaro JJ, McClure EA, Froeliger B. Effects of Hyperdirect Pathway Theta Burst Transcranial Magnetic Stimulation on Inhibitory Control, Craving, and Smoking in Adults With Nicotine Dependence: A Double-Blind, Randomized Crossover Trial. Biol Psychiatry Cogn Neurosci Neuroimaging. 2023 Nov;8(11):1156-1165. doi: 10.1016/j.bpsc.2023.07.014. Epub 2023 Aug 9. PMID 37567363

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 63 participants were consented and screened. 19 were excluded, 7 due to screen failure, 6 due to lost to follow up, 5 were participant initiated withdrawal and 1 due to investigator initiated withdrawal.
Pre-assignment Details: Of the 44 participants, 3 were excluded - 2 due to lost to follow up and 1 due to investigator initiated withdrawal. A total of 41 participants were randomized and started treatment.
Groups:
- Intermittent Theta-burst Stimulation (iTBS) First: Cross-over design - participants will receive both experimental treatments. Intermittent Theta-burst stimulation (iTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected.
  Continuous Theta-burst stimulation (cTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Continuous TBS (cTBS) which is thought to temporarily dampen brain activity in that specific area.
- Continuous Theta-burst Stimulation (cTBS) First: Cross-over design - participants will receive both experimental treatments. Continuous Theta-burst stimulation (cTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Continuous TBS (cTBS) which is thought to temporarily dampen brain activity in that specific area.
  Intermittent Theta-burst stimulation (iTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected.
Period: Second TBS
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) First | Continuous Theta-burst Stimulation (cTBS) First
Started | 20 | 21
Completed | 16 | 21
Not Completed | 4 | 0
Period: First TBS
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) First | Continuous Theta-burst Stimulation (cTBS) First
Started | 20 | 21
Completed | 16 | 21
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) First | Continuous Theta-burst Stimulation (cTBS) First | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 21 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 17 | 17 | 34
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: The Effects of cTBS vs. iTBS TMS Applied to the r.IFG on Change in Behavioral Inhibition Between Baseline and 1 Hour Post Treatment.
Description: Changes in errors of omission on an inhibitory control task performed prior to and immediately after cTBS, and changes in errors of omission on an inhibitory control task performed prior to and immediately after iTBS. Outcomes will be measured as the mean change in behavioral performance percent correct on inhibition trials between baseline and 1 hour post treatment. Scores on the inhibitory control task range from 0% correct to 100% correct, and the change from pre-post TBS is expressed as a percent increase or decrease in performance. Positive values represent an improved outcome, whereas negative values represent a worse outcome.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: Percentage of correct trials
Groups:
- Intermittent Theta-burst Stimulation (iTBS): Intermittent Theta-burst stimulation (iTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. The total duration of the iTBS protocol is 190 seconds. Participants will receive stimulation over the r.IFG (A series of 3-pulse bursts at 50 Hz repeated every 200ms (5 Hz) per train, 2 seconds per train, 20 trains, 10 second intertrain interval, 600 total pulses; 80% Resting Motor Threshold) using a figure 8 coil.
- Continuous Theta-burst Stimulation (cTBS): Continuous Theta-burst stimulation (cTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Continuous TBS (cTBS) which is thought to temporarily dampen brain activity in that specific area. The total duration of the cTBS protocol is 40 seconds. Participants will receive stimulation over the r.IFG (A series of 3-pulse bursts at 50 Hz repeated every 200 ms (5 Hz), 600 total pulses; 80% Resting Motor Threshold) using a figure 8 coil.
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) | Continuous Theta-burst Stimulation (cTBS)
Number analyzed (Participants) | 37 | 37
Percentage of correct trials | -3.078 (1.560) | 3.778 (2.006)

2. Primary Outcome: The Effects of cTBS vs. iTBS TMS Applied to the r.IFG on Changes in Craving to Smoke 1 Hour Post Treatment.
Description: Changes in self-reported craving to smoke will be assessed using the Questionnaire on Smoking Urges brief (QSUb) at 1 hour post session on each of three conditions (Baseline, cTBS, iTBS). The values are calculated as the mean of the scores between conditions at 1 hour post session. Scores on the QSUb range from 10 to 70. The lower the score, the better the outcome.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) | Continuous Theta-burst Stimulation (cTBS)
Number analyzed (Participants) | 32 | 32
Score on a scale | 37.281 (2.191) | 34.593 (2.547)

3. Primary Outcome: The Effects of cTBS vs. iTBS TMS Applied to the r.IFG on Changes in Craving to Smoke 24hrs Post Treatment Between Conditions.
Description: Changes in self-reported craving to smoke will be assessed using the Questionnaire on Smoking Urges brief (QSUb) at 24hrs post session on each of three conditions (Baseline, cTBS, iTBS). The values are calculated as the mean of the scores between conditions at 24 hours post session. Scores on the QSUb range from 10 to 70. The lower the score, the better the outcome.
Time Frame: 24 hours
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) | Continuous Theta-burst Stimulation (cTBS)
Number analyzed (Participants) | 32 | 32
Score on a scale | 28.656 (2.581) | 26.031 (2.071)

4. Primary Outcome: The Effects of cTBS vs. iTBS TMS Applied to the r.IFG on Changes in Craving to Smoke 48hrs Post Treatment Between Conditions.
Description: Changes in self-reported craving to smoke will be assessed using the Questionnaire on Smoking Urges brief (QSUb) at 48hrs post session on each of three conditions (Baseline, cTBS, iTBS). The values are calculated as the mean of the scores between conditions at 48 hours post session. Scores on the QSUb range from 10 to 70. The lower the score, the better the outcome.
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) | Continuous Theta-burst Stimulation (cTBS)
Number analyzed (Participants) | 32 | 32
Score on a scale | 29.781 (2.613) | 28.968 (2.275)

5. Primary Outcome: The Effects of cTBS vs. iTBS TMS Applied to the r.IFG on Changes in Hyperdirect Brain Circuit Function Between Pre and Post Session.
Description: Changes in inhibitory control task functional connectivity between the r.IFG and nodes within the hyperdirect pathway (r.SMA, r.STN) prior to and immediately after cTBS, and changes in inhibitory control task functional connectivity between the r.IFG and nodes within the hyperdirect pathway (r.SMA, r.STN) prior to and immediately after iTBS. Outcomes will be measured as the transformed correlation (rZ value) of BOLD functional connectivity collected during the inhibitory task. The higher the rZ, the better the outcome.
Time Frame: 1 hour
Measure: Mean (Standard Error); unit: Mean change in rz score.
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) | Continuous Theta-burst Stimulation (cTBS)
Number analyzed (Participants) | 37 | 37
Mean change in rz score. | -3.078 (1.56) | .321 (2.136)

ADVERSE EVENTS:
Time Frame: 48 hours post treatment for each condition - baseline, iTBS, cTBS
Groups:
- Intermittent Theta-burst Stimulation (iTBS): Intermittent Theta-burst stimulation (iTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected.The total duration of the iTBS protocol is 190 seconds. Participants will receive stimulation over the r.IFG (A series of 3-pulse bursts at 50 Hz repeated every 200ms (5 Hz) per train, 2 seconds per train, 20 trains, 10 second intertrain interval, 600 total pulses; 80% Resting Motor Threshold) using a figure 8 coil.
- Continuous Theta-burst Stimulation (cTBS): Continuous Theta-burst stimulation (cTBS): Theta-burst stimulation (TBS), a form of repetitive transcranial magnetic stimulation (rTMS), affects brain areas stimulated directly underneath the scalp and brain areas that are functionally connected. Continuous TBS (cTBS) which is thought to temporarily dampen brain activity in that specific area.The total duration of the cTBS protocol is 40 seconds. Participants will receive stimulation over the r.IFG (A series of 3-pulse bursts at 50 Hz repeated every 200 ms (5 Hz), 600 total pulses; 80% Resting Motor Threshold) using a figure 8 coil.
Arm/Group | Intermittent Theta-burst Stimulation (iTBS) | Continuous Theta-burst Stimulation (cTBS)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/37
Other Adverse Events (participants affected / at risk) | 8/41 | 8/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent Theta-burst Stimulation (iTBS) (N=41) | Continuous Theta-burst Stimulation (cTBS) (N=37)
Headache (Nervous system disorders) | 7 | 7
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 | 2
Arm/Hand Pain (General disorders) | 0 | 2
Numbness (Nervous system disorders) | 1 | 0
Weakness (Nervous system disorders) | 2 | 2
Loss of Dexterity (Nervous system disorders) | 1 | 1
Change in Vision (Eye disorders) | 0 | 1
Change in Hearing (Ear and labyrinth disorders) | 1 | 2
Tinnitis (Ear and labyrinth disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Loss of Appetite (Gastrointestinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT03960138/Prot_SAP_000.pdf